CLINICAL TRIAL: NCT05703399
Title: Long Term Followup of Patients Enrolled in MC1137 (BEAUTY)
Brief Title: Long Term Followup of Patients Enrolled in MC1137, BEAUTY Study
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC210301; NCI-2022-09616 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC210301 (Other: Mayo Clinic in Rochester); 21-010580 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-12-27; First posted 2023-01-30 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, questionnaire): Patients undergo collection of blood samples throughout the study. Patients may also complete questionnaires and undergo the collection of tissue samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and tissue samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This study gathers information and samples for further analysis as part of the BEAUTY study. The purpose of the BEAUTY study was to better understand the reasons why or why not breast cancers respond to standard chemotherapy. Collecting samples of blood and tissue and health and treatment information from patients on the BEAUTY study may help doctors identify changes that make cancer better respond to standard chemotherapy and develop better therapies for the treatment of cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the association of residual cancer burden and breast cancer disease-free interval.

II. Evaluate the trajectory of circulating tumor cell (CTC) and circulating tumor-deoxyribonucleic acid (ctDNA) over time after breast cancer treatment and the association with breast cancer disease-free interval.

III. Evaluate the association of peripheral blood immune phenotype (circulating immune cell subpopulations as measured by cytometry by time-of-flight [CyTOF]) over time with breast cancer disease-free interval.

IV. Develop and use patient derived xenograft (PDX) models from recurrent breast cancer to identify mechanisms of treatment resistance and to study new drugs/drug combinations.

V. Evaluate changes in the genomic and proteomic landscape over time, by sequencing recurrent disease and comparing with sequencing data from the primary tumor.

VI. Assess the spatial immune micro-landscapes of pre-treatment and treated tumors.

VII. Generate autologous co-culture systems of peripheral blood immune cells and breast cancer tumor cells to study the endogenous antitumor immune response and immune evasion mechanisms.

OUTLINE:

Patients undergo collection of blood samples throughout the study. Patients may also complete questionnaires and/or undergo the collection of tissue samples throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION - FOR PATIENTS STILL ALIVE:
* Enrolled in BEAUTY [MC1137 (NCT02022202)] and did not withdraw consent while enrolled on BEAUTY for either specimen collection or long-term follow-up
* Able to provide written informed consent
* REGISTRATION - FOR PATIENTS WHO HAVE DIED:
* Enrolled in MC1137 and did not withdraw consent while enrolled on BEAUTY for either specimen collection or long-term follow-up
* Existence of a family member willing to provide consent for use of archived tumor biopsies obtained after enrollment in BEAUTY

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled in BEAUTY (MC1137) and did not withdraw consent while enrolled on BEAUTY for either specimen collection or long-term follow-up
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Association of residual cancer burden and breast cancer disease-free interval | Up to 10 years following study entry
Trajectory of CTC and ctDNA over time after breast cancer treatment | Up to 10 years following study entry
  Using RareCyte CTC technology
Association with breast cancer disease-free interval | Up to 10 years following study entry
Association of peripheral blood immune phenotype (circulating immune cell subpopulations as measured by CyTOF) over time with breast cancer disease-free interval | Up to 10 years following study entry
Identification of mechanisms of treatment resistance and to study new drugs/drug combinations | Up to 10 years following study entry
  Will develop and use PDX models from recurrent breast cancer to identify mechanisms of treatment resistance and to study new drugs/drug combinations.
Changes in the genomic and proteomic landscape over time | Up to 10 years following study entry
  Will evaluate changes in the genomic and proteomic landscape over time, by sequencing recurrent disease and comparing with sequencing data from the primary tumor.
Assess Spatial immune micro-landscapes of pre-treatment and treated tumors | Up to 10 years following study entry
  High-plex digital spatial profiling will be used to evaluate immune biomarkers
Endogenous antitumor immune response and immune evasion mechanisms | Up to 10 years following study entry
  Will generate autologous co-culture systems of peripheral blood immune cells and breast cancer tumor cells to study the endogenous antitumor immune response and immune evasion mechanisms

CONTACTS AND LOCATIONS:
Overall Officials: Judy C. Boughey, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials